CLINICAL TRIAL: NCT05998876
Title: Assessing Dose Taken in Opioid Use Disordered Patients With an Electrochemical Sensor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cari Health Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IRB005
Record Dates: First submitted 2023-08-06; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Adherence, Medication; Opioid Use Disorder
Keywords: Pharmacokinetics; Differential Pulse Voltammetry; Remote Medication Monitor; Interstitial Fluid
MeSH Terms: conditions — Medication Adherence; Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- 3-6 HRS: Microneedle electrode array placed into dermis for up to 6 hours. DPV Scans performed at a frequency of 1-20 per hour.
  Interventions: Device: Remote Medication Monitor (RMM) - Prototype; Drug: Daily Methadone Dose
- 12 HRS: Microneedle electrode array placed into dermis for up to 12 hrs. DPV Scans performed at a frequency of 1-20 per hour.
  Interventions: Device: Remote Medication Monitor (RMM) - Prototype; Drug: Daily Methadone Dose
- 3 Days: Microneedle electrode array placed into dermis for up to 3 days. DPV Scans performed at a frequency of 1-20 per hour.
  Interventions: Device: Remote Medication Monitor (RMM) - Prototype; Drug: Daily Methadone Dose

INTERVENTIONS:
Device: Remote Medication Monitor (RMM) - Prototype — Inserted Microneedle Electrode Array for assaying dermal interstitial fluid.
  Other Names: RMM
Drug: Daily Methadone Dose — patient takes their prescribed daily dose of methadone
  Other Names: Dose Taken

SUMMARY:
CARI Health aims to develop a methadone dose taken sensor that provides real-time data on interstitial fluid (ISF) levels that could be used as a methadone adherence monitor for daily doses. Use of such a monitor would allow for the physician, counselor, patient, and family member to remotely verify that a physician prescribed dose has been taken. Such a verification system can allow methadone clinics greater flexibility in the provision of take-home doses and thus retain more patients in the clinic.

DETAILED DESCRIPTION:
Three specific phases and 9 aims are proposed for first-in-human studies of a remote medication monitor for dose taken in patients taking methadone for opiate use disorder.

Phase 1 detection over 3-6 hours (N=10)

Aim 1: Detect methadone and one or more of its metabolites in interstitial fluid (ISF) with differential pulse voltammetry (DPV) Aim 2: Correlate in vitro blood-based LC-MS and DPV Scans with Intradermal Microneedle based DPV Scans Aim 3: Accurately identify that a dose of methadone has been taken Aim 4: Determine the frequency and severity of any adverse events up to 6 hours.

Phase 2 detection over 12 hours (N=15)

Aim 5. Quantitate methadone and one or more of its metabolites in ISF with DPV over 12 hrs.

Aim 6: Determine the frequency and severity of any adverse events up to 12 hours

Phase 3 detection over 3 days N=20 ( 15 single dosed subjects, 5 split dosed subjects )

Aim 7. Quantitate methadone and one or more of its metabolites in ISF with DPV over 3 days.

Aim 8. Accurately identify a dose or half a dose has been taken Aim 9: Determine the frequency and severity of any adverse events up to 3 days

ELIGIBILITY:
Inclusion criteria for methadone group includes:

Age 18-70. A prescription for liquid methadone at a dose of 10mg or more. Taken methadone as prescribed in the last 2 days. Has been prescribed at least 3 take homes

Exclusion criteria for methadone group includes:

Age <18 or >70. A condition preventing or complicating ISF collection. Conditions may include dermatological (skin) condition, immunodeficiency, bleeding diathesis, recent blood donation, anemia, cancer, congestive heart failure, or tuberculosis. Any active severe depression (e.g., suicidal ideation) or mania symptoms.

Pregnancy, or intending to become pregnant during the course of the study. Patients determined to be unstable for enrollment or take homes by the Outpatient Treatment Program (OTP).

Under a conservatorship.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients taking methadone for opioid use disorder
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of detection of methadone levels in Interstitial Fluid using an electrochemical sensor | from 3 hours to 3 days.
  Sensitivity of Repeated measurements of methadone levels
Specificity of detection of methadone levels in Interstitial Fluid using an electrochemical sensor | from 3 hours to 3 days.
  Specificity of Repeated measurements of methadone levels

SECONDARY OUTCOMES:
Correlation between Blood and ISF levels of Methadone and Methadone Metabolites assayed with Liquid Chromatography - Mass Spectroscopy (LC-MS) | from 3 hours to 3 days
  Pearson coefficient
Correlation between Blood and ISF levels of Methadone and Methadone Metabolites assayed with Remote Medication Monitor | from 3 hours to 3 days
  Pearson coefficient
Correlation between Liquid Chromatography - Mass Spectroscopy (LC-MS) and Differential Pulse Voltammetry (DPV) | from 3 hours to 3 days
  Pearson Coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Bari, MD, Principal Investigator — Synergy Research Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Cari Health Website — http://www.carihealth.com